CLINICAL TRIAL: NCT03129321
Title: Clinical Study to Evaluate the Therapeutic Equivalence and Safety of Econazole Nitrate Cream, 1% (Renaissance Pharma, Inc.) to Econazole Nitrate Cream, 1% (Perrigo New York Inc.) in Tinea Pedis
Brief Title: Therapeutic Equivalence and Safety of Two Econazole Nitrate Cream, 1% Products in Tinea Pedis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: DPT Laboratories, Ltd. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 71532902
Record Dates: First submitted 2017-04-05; First posted 2017-04-26 (Actual); Results first posted 2018-08-02 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Tinea Pedis
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Test (Experimental): Econazole Nitrate Cream, 1%, topical, sufficient amount to cover all affected areas on the feet once daily for 28 days
  Interventions: Drug: Econazole Nitrate Cream, 1%
- Reference Standard (Active Comparator): Econazole Nitrate Cream, 1%, topical, sufficient amount to cover all affected areas on the feet once daily for 28 days
  Interventions: Drug: Econazole Nitrate Cream, 1%
- Placebo (Placebo Comparator): Placebo Cream, topical, sufficient amount to cover all affected areas on the feet once daily for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Econazole Nitrate Cream, 1%
  Arms: Reference Standard; Test
Drug: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the therapeutic equivalence of the Test formulation, econazole nitrate cream, 1% to the Reference product, econazole nitrate cream, 1% in the treatment of tinea pedis.

To demonstrate the superiority of the Test and Reference (active) treatments over Placebo treatment in patients with tinea pedis.

To compare the safety of Test, Reference and Placebo treatments in patients with tinea pedis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant, non-lactating female ≥ 18 years of age.
* Clinical diagnosis of tinea pedis with lesions localized to the interdigital spaces or predominantly interdigital, but may extend to other areas of the foot (the non-interdigital lesions should not be hyperkeratotic, i.e., characteristic of tinea pedis moccasin).
* Provisionally confirmed at baseline by a positive potassium hydroxide (KOH) wet mount preparation
* Total score ≥ 4 for the clinical signs and symptoms of tinea pedis in the target area. In addition the target area must have a minimum score of at least 2 for erythema and a minimum score of at least 2 for either pruritus or scaling.

Exclusion Criteria:

* Presence of any other infection of the foot or other disease process that, in the Investigator's opinion, may interfere with the evaluation of the patient's tinea pedis
* History of or current psoriasis, Lichen planus or contact dermatitis involving the feet within the previous 12 months.
* Past history of dermatophyte infections with a lack of response to antifungal therapy
* Confluent, diffuse moccasin-type tinea pedis of the entire plantar surface or onychomycosis involving ≥ 20% of the area of either great toenail and/or involving more than five toenails in total or other concurrent dermatophytoses (e.g., tinea cruris) and any other skin disease to an extent that, in the opinion of the investigator, might interfere with the evaluation of tinea pedis or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 876 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2016-11-17 (Actual); Study Completion 2016-11-17 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Test; Reference Standard: Econazole Nitrate Cream, 1%, topical, sufficient amount to cover all affected areas on the feet once daily for 28 days
  Econazole Nitrate Cream, 1%
- Placebo: Placebo Cream, topical, sufficient amount to cover all affected areas on the feet once daily for 28 days
  Placebo
Period: Overall Study
Arm/Group | Test | Reference Standard | Placebo
Started | 351 | 350 | 175
Completed | 253 | 241 | 120
Not Completed | 98 | 109 | 55

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test | Reference Standard | Placebo | Total
Number analyzed (Participants) | 351 | 350 | 175 | 876
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (12.9) | 47.1 (14.6) | 46.1 (13.3) | 47.0 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 114 | 60 | 301
  Male | 224 | 236 | 115 | 575
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 168 | 165 | 81 | 414
  Not Hispanic or Latino | 183 | 185 | 94 | 462
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 191 | 197 | 93 | 481
  Black/African American | 149 | 142 | 74 | 365
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 1
  Asian | 3 | 4 | 2 | 9
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Other | 7 | 6 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients in Each Active Treatment Group Who Are Considered a Therapeutic Cure
Description: To be considered a Therapeutic Cure, the patient must have both Clinical Cure (patient's total severity score must be ≤ 2 with no individual severity score > 1) and Mycological Cure (patient must have a negative KOH test and a negative fungal culture) of tinea pedis
Time Frame: Day 42
Population: Active Treatments of the Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Test | Reference Standard
Number analyzed (Participants) | 185 | 170
Participants | 96 | 81
Statistical Analysis 1: Comparison: Test vs Reference Standard; Test type: Equivalence — Equivalence margin: +/-20%; Difference in proportions = 4.24, 90% CI 2-sided [-5.05 to 13.54]

2. Primary Outcome: Proportion of Patients in Each Treatment Group Who Are Considered a Therapeutic Cure
Description: as for outcome 1
Time Frame: Day 42
Population: Modified Intent to Treat. Patients who are missing mycological culture data at baseline are not included in the analysis. Patients who are missing mycological culture data at the test of cure visit are not included in the analysis unless they were a treatment failure.
Measure: Count of Participants; unit: Participants
Arm/Group | Test | Reference Standard | Placebo
Number analyzed (Participants) | 201 | 188 | 90
Participants | 102 | 88 | 22
Statistical Analysis 1: Comparison: Test vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Reference Standard vs Placebo; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel

3. Secondary Outcome: Proportion of Patients in Each Active Treatment Group Who Are Considered a Clinical Cure (Patient's Total Severity Score Must be ≤ 2 With no Individual Severity Score > 1)
Description: The following Clinical Signs and Symptoms of a target lesion with tinea pedis are individually rated for severity (none, mild, moderate, or severe): fissuring/cracking, erythema, maceration, scaling, pruritus, and burning/stinging
Time Frame: Day 42
Population: Active treatment groups of the Per Protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Test | Reference Standard
Number analyzed (Participants) | 185 | 170
Participants | 113 | 99
Statistical Analysis 1: Comparison: Test vs Reference Standard; Test type: Equivalence — Equivalence margin: +/-20%; Difference in proportions = 2.85, 90% CI 2-sided [-6.29 to 11.98]

4. Secondary Outcome: Proportion of Patients in Each Active Treatment Group Who Are Considered a Mycological Cure
Description: To be considered a mycological cure the patient must have a negative KOH test and a negative fungal culture for T. rubrum, T. mentagrophytes or E. floccosum
Time Frame: Day 42
Population: Active treatment groups of the Per Protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Test | Reference Standard
Number analyzed (Participants) | 185 | 170
Participants | 136 | 125
Statistical Analysis 1: Comparison: Test vs Reference Standard; Test type: Equivalence — Equivalence margin: +/-20%; Difference in proportions = -0.02, 90% CI 2-sided [-8.29 to 8.26]

5. Secondary Outcome: Proportion of Patients in Each Treatment Group Who Are Considered a Clinical Cure (Patient's Total Severity Score Must be ≤ 2 With no Individual Severity Score > 1)
Description: as for outcome 3
Time Frame: Day 42
Population: Modified Intent to Treat
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo Cream, topical,
Arm/Group | Test | Reference Standard | Placebo
Number analyzed (Participants) | 214 | 198 | 95
Participants | 131 | 113 | 40
Statistical Analysis 1: Comparison: Test vs Placebo; Test type: Superiority; p = 0.0020, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Reference Standard vs Placebo; Test type: Superiority; p = 0.0076, Cochran-Mantel-Haenszel

6. Secondary Outcome: Proportion of Patients in Each Treatment Group Who Are Considered a Mycological Cure
Description: as for outcome 4
Time Frame: Day 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo Cream, topical, sufficient amount to cover all affected areas on the feet once daily for 28 days
  Placebo Cream
Arm/Group | Test | Reference Standard | Placebo
Number analyzed (Participants) | 201 | 188 | 90
Participants | 147 | 137 | 37
Statistical Analysis 1: Comparison: Test vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Reference Standard vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Arm/Group | Test | Reference Standard | Placebo
Serious Adverse Events (participants affected / at risk) | 0/351 | 0/350 | 0/175
Other Adverse Events (participants affected / at risk) | 0/351 | 0/350 | 0/175

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall not publish, or seek to publish, either in whole or in part any results of the study without the written consent of CRO.